CLINICAL TRIAL: NCT07068243
Title: Transverse Versus Longitudinal Approaches for Rectus Sheath Block: a Randomized Controlled Trial in Healthy Volunteers
Brief Title: REctus Sheath Trial
Acronym: REST
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00118293
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Pain; Postoperative Pain, Acute
Keywords: Rectus Sheath Block; Abdominal Block; Fascial Plane Block; RSB
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Transverse Approach to the Rectus Sheath Block (Active Comparator): In the transverse approach, the US probe will be positioned perpendicular to the he rectus abdominis muscle's fibers, and the needle will be inserted in-plane from lateral to medial.
  Interventions: Drug: 1.0% lidocaine with epinephrine (1:100,000)
- Longitudinal Approach to the Rectus Sheath Block (Experimental): In contrast, the longitudinal approach will involve aligning the probe parallel to the rectus muscle fibers, with the needle advanced in-plane from cephalad to caudad.
  Interventions: Drug: 1.0% lidocaine with epinephrine (1:100,000)

INTERVENTIONS:
Drug: 1.0% lidocaine with epinephrine (1:100,000) — The block will be performed by advancing the needle into the posterior rectus sheath compartment, with the local anesthetic deposited posterior to the rectus abdominis muscle and anterior to the posterior rectus sheath.
  Drug: 20 mL injection of 1.0% lidocaine with epinephrine (1:100,000) on each side (40mL total/subject)

SUMMARY:
Regional anesthesia techniques (or nerve blocks) are used to provide sensory blockade over the abdominal wall. The most established technique is thoracic epidural. This provides bilateral spread but is also associated with neuraxial complications, which has led to a decrease in clinical usage. The rectus sheath block (RSB) is an established regional anesthesia technique used to provide somatic analgesia to the midline anterior abdominal wall by depositing local anesthetic in the posterior rectus sheath, thereby targeting the terminal anterior branches of the lower thoracic intercostal nerves. The conventional approach involves placing the ultrasound (US) probe transversely across the rectus abdominis muscle and advancing the needle in-plane either lateral-to-medial or medial-to-lateral. While this technique achieves spread within the sheath, the cephalocaudal distribution of local anesthetic may be suboptimal, potentially limiting the extent of dermatomal coverage. A longitudinal probe orientation, with needle insertion from cephalad to caudad, may theoretically facilitate a more extensive cranio-caudal spread by aligning the injection axis with the anatomical fascial plane of the posterior rectus sheath. However, the relative efficacy of these two approaches has not been investigated in a controlled, comparative setting. Thus, this randomized, single-blinded trial aims to evaluate the dermatomal sensory distribution and ultrasound-assessed local anesthetic spread achieved by the transverse versus longitudinal in-plane approaches to ultrasound-guided RSB in healthy adult volunteers. To compare the dermatomal sensory block distribution, investigators will use dermatomal mapping with pinprick, and cold.

DETAILED DESCRIPTION:
A total of 14-18 adult volunteers will be included. Each participant will receive bilateral rectus sheath blocks at a standardized supraumbilical level. The side receiving the transverse approach (US probe perpendicular to muscle fibers; needle in-plane lateral-to-medial) and the side receiving the longitudinal approach (US probe parallel to muscle fibers; needle in-plane cephalad-to-caudad) will be randomized. The blocks will be performed with a standardized volume and concentration of local anesthetic, under real-time US guidance by the same experienced anesthesiologist. The research team member assessing the block will be blinded. Immediately after injection of each block, US imaging will be used to assess and measure the length and pattern of spread within the posterior rectus sheath. At baseline and at 60 minutes post-block, dermatomal sensory mapping will be performed using standardized cold and pinprick stimuli over the anterior abdominal wall.

ELIGIBILITY:
Inclusion criteria:

1. Ability to provide written informed consent
2. Ability and willingness to comply with the study procedures and duration requirements
3. ASA physical status 1 or 2
4. Age ≥ 18 years
5. Weight > 60kg

Exclusion criteria:

1. BMI > 40kg.m-2
2. Use of analgesics within 24 hours before the procedure
3. History of abdominal trauma or surgery
4. Abdominal deformities or abnormalities that may prevent proper block performance
5. Abdominal tattoos in the supraumbilical area
6. Systemic neuromuscular disease
7. Contraindications to regional anesthesia (e.g., infection, allergy)
8. Structures are unable to be visualized by ultrasound
9. Pregnancy
10. Other known health conditions that would affect the participant's ability to successfully complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Temperature discrimination | 60 to 90 minutes post-block
  Skin temperature assessment using gloved ice on the chest wall, to discriminate blocked vs unblock areas.
Mechanical discrimination | 60 to 90 minutes post-block
  Mechanical assessment using a neuropin (pinprick) on the chest wall, to discriminate blocked vs unblock areas.
Cutaneous distribution mapping | 60 to 90 minutes post-block
  Mapping the blocked area (using the previous temperature and mechanical assessments, demarcating lines on the skin) to provide a visual map and, to calculate the area blocked.

SECONDARY OUTCOMES:
Direct visualization of the local anesthetic spread | Immediately post-block
  Direct visualization of the local anesthetic spread cephalad and caudad, marking the highest and lowest dermatomes where local anesthetic was still seen on the US, with the US oriented longitudinally.
Measurement of the local anesthetic spread in each dermatome with the US | Immediately post-block
  Measurement of the local anesthetic spread in each dermatome with the US oriented transversely, by measuring hypoecoic area produced by the presence of local anesthetic.

OTHER OUTCOMES:
Adverse Events | End of study (2 days post blocks).
  Any adverse events block-related will be recorded

IPD SHARING:
Plan to Share IPD: No